CLINICAL TRIAL: NCT05952492
Title: Improving Young Adult Cancer Survivors' Mental Health with an EHealth Group Intervention
Brief Title: Digital Connections: an EHealth Group Intervention for Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003230
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stress Management Skills Training (Experimental): Participants will attend group sessions with a trained facilitator held over videoconference. Sessions will each last 2 hours and be held once weekly for 10 weeks. Sessions will include stress management skills training and health education content.
  Interventions: Behavioral: Stress Management Skills Training

INTERVENTIONS:
Behavioral: Stress Management Skills Training — Participants will attend group sessions with a trained facilitator held over videoconference. Sessions will each last 2 hours and be held once weekly for 10 weeks. Sessions will include stress management skills training and health education content.

SUMMARY:
The purpose of this study is to determine the feasibility of recruiting young adult cancer survivors from across the nation and to explore the impact of an eHealth group intervention on psychosocial health in this population.

DETAILED DESCRIPTION:
Study investigators will conduct a single-arm pilot trial in which a 10 week eHealth group intervention will be delivered via a study website. We will use a multi-pronged approach to recruit young adult cancer survivors from across the country. Study participants will attend weekly group meetings with a trained facilitator to receive the manualized intervention over the course of 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-39 years at the time of participation
2. Diagnosed with any invasive cancer between 15-39 years old
3. Finished curative cancer treatment 1 month to 5 years prior to enrollment (except maintenance therapy such as ongoing hormone therapy)
4. Currently experiencing at least mild symptoms of depression or anxiety (i.e., score ≥1 on the Patient Health Questionnaire-4)
5. Able to speak and read English so all group attendees can communicate in a shared language.
6. Able and willing to give informed consent.
7. Access to internet or cellular connectivity with sufficient bandwidth to participate in videoconferences

Exclusion Criteria:

1) Documented or observable psychiatric or neurological disorders that could interfere with study participation (e.g., psychosis, active substance abuse)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment of young adult cancer survivors | Through study completion, an average of 1 year
  Recruitment will be considered feasible if ≥40% of eligible survivors enroll in the study.

SECONDARY OUTCOMES:
Change in health-related quality of life from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the 27-item Functional Assessment of Cancer Therapy - General. Scores range from 0 to 108, with higher scores reflecting better quality of life.
Change in stress management self-efficacy skills from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete subscales from the Measure of Current Status. Subscale scores range from 0 to 8, 0 to 12, or 0 to 20 depending on the subscale. Higher scores indicate more of the construct being assessed.
Change in cancer-related distress from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the 22-item Impact of Event Scale-Revised. Scores range from 0 to 88, with higher scores indicating greater cancer-related distress.
Change in coping from baseline to immediately after the intervention | Baseline and immediately after the intervention
  Participants will complete the Brief Coping Orientation to Problems Experienced scale, which yields 14 two-item subscales. Subscale scores range from 2 to 8, with higher scores indicating greater usage of the coping strategy being assessed.
Change in anxiety symptoms from baseline to immediately after the intervention | Baseline and immediately after the intervention.
  Participants will complete the Generalized Anxiety Disorder-7. Given the sample size, the investigators will focus on effect sizes rather than statistical significance.
  The Unabbreviated scale title is the Generalized Anxiety Disorder-6. Minimum value=0. Maximum value=21. Higher scores=worse.
Change in depression symptoms from baseline to immediately after the intervention | Baseline and immediately after the intervention.
  Participants will complete the Patient Health Questionnaire-9. Given the sample size, the investigators will focus on effect sizes rather than statistical significance.
  The Unabbreviated scale title is the Patient Health Questionnaire-9. Minimum value=0. Maximum value=27. Higher scores=worse.
Change in trend and relative values of time and frequency domain heart rate variability metrics from pre- to post-intervention. | Baseline and the final week of the intervention
  Participants will wear a wearable sensor for at least 1 week.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Fox, PhD, MPH, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fox RS, Badger TA, Moya S, Gudenkauf LM, Nelson MA, O'Neill RM, Leete JJ, Friedman SE, Katsanis E, Victorson DE, Sanford SD, Penedo FJ, Antoni MH, Oswald LB. An HRQOL Proof-Of-Concept Analysis of the eHealth TOGETHER Intervention for Adolescent and Young Adult Cancer Survivors: A Brief Report. Psychooncology. 2025 Jul;34(7):e70234. doi: 10.1002/pon.70234. PMID 40879639